CLINICAL TRIAL: NCT03588728
Title: tDCS and Cognitive Training Intervention for Chronic Smokers With Schizophrenia
Acronym: TACTICSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lab was shut down due to COVID as were nearing study completion
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Cynthia Conklin, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS; R21DA045137 (NIH)
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-12

CONDITIONS: Transcranial Direct Current Stimulation; Smoking, Cigarette; Schizophrenia
Keywords: Transcranial Direct Current Stimulation; Smoking; Schizophrenia
MeSH Terms: conditions — Cigarette Smoking; Schizophrenia; Smoking | interventions — Transcranial Direct Current Stimulation; Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: 2 (CR, Control CR) x 2 (tDCS xSham tDCS)
Who Masked: Participant
Masking Description: Participants were not informed of their randomization group until debreifing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CR + tDCS (Experimental): Cognitive Remediation (CR) and Transcranial Direct Current Stimulation (tDCS)
  Interventions: Other: Transcranial Direct Current Stimulation; Behavioral: Cognitive Remediation (CR)
- CR + sham tDCS (Sham Comparator): Cognitive Remediation (CR) and Sham Transcranial Direct Current Stimulation (tDCS)
  Interventions: Behavioral: Cognitive Remediation (CR)
- control CR + tDCS (Sham Comparator): Control Cognitive Remediation (CR) and Transcranial Direct Current Stimulation (tDCS)
  Interventions: Other: Transcranial Direct Current Stimulation
- control CR + sham tDCS (No Intervention): Control Cognitive Remediation (CR) and Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — Transcranial direct current stimulation targeting the right inferior frontal gyrus
  Other Names: tDCS
  Arms: CR + tDCS; control CR + tDCS
Behavioral: Cognitive Remediation (CR) — Cognitive exercises on a computer designed to increase attention, memory, and processing speed.
  Arms: CR + sham tDCS; CR + tDCS

SUMMARY:
This study is being done to develop new methods to help smokers with schizophrenia to successfully reduce their smoking and/or quit. This is not a treatment study, but will help find new techniques to create better treatments. Specifically, the investigators are interested in learning more about how thoughts and attention problems associated with schizophrenia might play a role in smoking, as well as the impact of cognitive (thinking, reasoning, and remembering) training and brain stimulation on these symptoms and on actual smoking.

DETAILED DESCRIPTION:
Adults with severe mental illness (SMI) are three times more likely to smoke than non-SMI adults, consuming 35-44% of all cigarettes in the U.S.; and, the highest rates of tobacco-related illnesses and death are among smokers with schizophrenia. Unfortunately, not only are patients with schizophrenia less likely to receive smoking treatments, but cessation medications are only modestly effective in helping this subset of smokers quit. Therefore, it is vital to discover new treatment adjuncts that specifically aid this high-risk subset of smokers to achieve successful abstinence. Toward that end, the investigators propose a novel non-pharmacologic technique that directly targets both cognitive impairment, an avenue considerable past research suggests may be particularly effective to exploit in smokers with schizophrenia, and reactivity to prepotent stimuli, shown to be enhanced in smokers with schizophrenia. Combining a subset of cognitive enhancement therapy known as Cognitive Remediation (CR), with another safe and effective technique, Transcranial Direct Current Stimulation (tDCS), the investigators propose a new cognitive training method aimed at enabling smokers with schizophrenia to gain greater control over smoking and stimuli-induced reactivity (e.g., craving). Recent studies have found significant tDCS-induced cognitive enhancement, as well as reduction in both cue-induced craving and smoking behavior among healthy smokers. This combined with knowledge of the cognitive deficits that exist among individuals with schizophrenia, and clear evidence of a relationship between cognitive function and smoking treatment success, provides the rationale for testing novel CR + tDCS to target underlying mechanisms of smoking among individuals with schizophrenia. Specifically, the proposed study will examine the extent to which targeted cognitive enhancement with CR + tDCS, leads to changes in cognitive control, cue-provoked craving, reaction time and ERP measures of attentional bias; as well as the impact of these changes on smoking behavior and intention and confidence to quit among 80 smokers with schizophrenia. The goal of this study is to inform the development of new non-medication, noninvasive, therapeutic techniques to specifically target smoking among patients with schizophrenia. The long term goal is to establish an effective treatment adjunct to help smokers with schizophrenia successfully achieve abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Currently meets DSM-5 criteria for Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder, or Delusional Disorder.
* Ability to provide written informed consent
* Smoke ≥ 7 cigarettes per day
* Expired breath CO ≥ 10 ppm at screening
* Stable medication regimen for ≥ 4 weeks (If on more than one psychotropic medication, main antipsychotic will be considered for stability)

Exclusion Criteria:

* Epilepsy or Current Seizure Disorder
* Alcohol or Substance Dependence past 3 months (caffeine allowed, nicotine is part of inclusion criteria).
* Pregnant or lactating
* Psychiatric hospitalization in past 3 months
* Suicidal and/or aggressive behavior past 3 months
* Implanted cardiac or brain medical devices
* Latex allergy
* Scalp irritation or recent shaving of scalp
* Use of other smoking cessation medication
* History of head trauma
* History of ECT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Conklin, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Started | 10 | 6 | 12 | 11
Completed | 7 | 6 | 9 | 8
Not Completed | 3 | 0 | 3 | 3
Not completed — Did not meet eligibility ctriteria | 0 | 0 | 3 | 2
Not completed — Lab shut down due to COVID-19 | 0 | 0 | 0 | 1
Not completed — multiple technical issues | 1 | 0 | 0 | 0
Not completed — Hospitalized for COVID | 1 | 0 | 0 | 0
Not completed — Schedule change unable to attend sessions | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: These number reflect participants who completed the study. 3 of 10 participants in CR + tDCS did not complete. 3 of 12 participants in control + tDCS did not complete. 3 of 11 participants in CR + tDCS did not complete. Total from Study Flow = 39 with 30 Completers
Groups:
- Total: Total of all reporting groups
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS | Total
Number analyzed (Participants) | 7 | 6 | 9 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 9 | 8 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (13.0) | 52.5 (9.4) | 50.9 (8.3) | 48.4 (10.5) | 49.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 2 | 12
  Male | 5 | 2 | 5 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 8 | 7 | 26
  Unknown or Not Reported | 2 | 0 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 5 | 17
  White | 3 | 1 | 4 | 3 | 11
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 9 | 8 | 30
Nicotine Dependence Score [Mean (Standard Deviation); unit: units on a scale] — Level of dependence measured 0-7 with a higher score indicating more nicotine dependence.
  units on a scale | 4.7 (1.7) | 5.8 (1.6) | 5.0 (1.1) | 5.8 (2.0) | 5.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS™): MATRICS Consensus Cognitive Battery (MCCB)
Description: the MATRICS Consensus battery (MCCB) is a cognitive battery of tests for assessing cognition-enhancing treatments for schizophrenia through a broadly based scientific evaluation of measures. Change in cognitive measures of MATRICS Consensus Cognitive Battery (MCCB). Post-intervention minus baseline. Scale is scored 0-100. Difference score range is (-100 to 100) with positive scores reflecting improvement.
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 7 | 6 | 9 | 8
score on a scale | 3.6 (4.0) | 2.3 (8.6) | 3.1 (3.6) | 1.8 (3.7)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-subjects effects; Test type: Superiority; p = .781, ANOVA; P value indicates the interaction term

2. Secondary Outcome: Cue-Reactivity
Description: Change in cue-induced craving indexed as change in self-report craving on the questionnaire of smoking urges, 4-item version (QSU-4) from baseline to end of intervention. Craving rating range = 0-100. Difference scores range from (-100 to 100) with a negative score reflecting improvement.
Time Frame: Baseline to approximately 4 weeks
Population: Three subjects were removed from analyses due to misunderstanding the computerized rating system.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 6 | 5 | 9 | 7
score on a scale | -6.4 (38.1) | -6.2 (14.3) | -3.0 (24.5) | 2.6 (29.5)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-subjects effects; Test type: Superiority; p = .409, ANOVA; P value indicates the interaction term

3. Secondary Outcome: Cigarette Puff Volume
Description: Change in mean cigarette puff volume
Time Frame: Baseline and at approximately 4 weeks
Population: Participants who did not smoke at baseline during cue reactivity were excluded from the analyses. This included 1 from arm CR + tDCS, 2 from CR + sham tDCS, and 2 from control CR + tDCS.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 6 | 4 | 7 | 8
Milliliters | -218.8 (450.9) | -90.7 (345.0) | -9.9 (268.0) | 27.4 (623.5)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-subjects effects; Test type: Superiority; p = .697, ANOVA; P value indicates the interaction term

4. Secondary Outcome: Latency to First Cigarette Puff
Description: Change in mean latency to first cigarette puff
Time Frame: Baseline to approximately 4 weeks
Population: Participants who did not smoke at baseline during cue reactivity were excluded from this analysis. This included 1 from arm CR + tDCS, 2 from CR + sham tDCS, and 2 from control CR + tDCS.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 6 | 4 | 7 | 8
seconds | 119.0 (197.1) | 182.8 (243.7) | 19.1 (65.1) | 96.5 (188.3)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between subjects effects; Test type: Superiority; p = .193, ANOVA; P value indicates interaction term

5. Secondary Outcome: AX Version of the Continuous Performance Task (AX-CPT) Reaction Time
Description: AX version of the CPT measures a participant's active maintenance and cognitive control. In this task, the participant is presented with a series of trials in which they are instructed to make a response which distinguishes between stimuli. Here the stimuli included are: smoking, nonsmoking, person, non-person). Assessment is of Post - Pre intervention difference in reaction time to respond to stimuli on the AX Version of the Continuous Performance Task (AX-CPT)
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 7 | 6 | 9 | 8
milliseconds | -59.5 (62.9) | -37.8 (47.4) | 4.3 (29.8) | -7.2 (30.8)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-subjects effects; Test type: Superiority; p = .185, ANOVA; P value indicates the interaction term

6. Secondary Outcome: AX Version of the Continuous Performance Task (AX-CPT) Reaction Time Variability
Description: Post minus pre-intervention difference Reaction time variability for hits on the AX Version of the Continuous Performance Task (AX-CPT). A negative value indicates improvement.
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 7 | 6 | 9 | 8
milliseconds | -49463.5 (71684.1) | 12828.3 (63752.7) | 22570.7 (83194.9) | 8292.96 (74462.3)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-measures effects; Test type: Superiority; p = .198, ANOVA; P value indicates the interaction term

7. Secondary Outcome: EEG (Electroencephalogram) N170 Amplitude
Description: Difference in change scores (post minus pre-intervention) in N170 Amplitude between smoking and neutral images. A more negative score indicates greater improvement.
Time Frame: Baseline to approximately 4 weeks
Population: Subjects were removed from analysis if their data was too noisy from excessive coughing or moving around.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 7 | 5 | 6 | 5
microvolts | -1.9 (1.8) | 0.2 (1.9) | -0.8 (2.2) | 0.6 (1.3)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-subjects effects; Test type: Superiority; p = .638, ANOVA

8. Secondary Outcome: EEG (Electroencephalogram) Contingent Negative Variation (CNV)
Description: Difference in CNV between the A and X in the AX-CPT Task. More negative indicates larger CNV.
Time Frame: Baseline to approximately 4 weeks
Population: Subjects were removed from analysis if their data was too noisy from excessive coughing or moving around.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 7 | 5 | 7 | 5
microvolts | 0.8 (1.7) | 0.6 (1.5) | 0.8 (1.3) | 1.2 (1.1)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-subjects effectd; Test type: Superiority; p = .574, ANOVA; p-value indicates the interaction term

9. Secondary Outcome: EEG (Electroencephalogram) Beta-Band Event-Related Desynchronization (ERD)
Description: Difference in ERD between the A and X in AX-CPT during EEG assessment of Beta-Band Event-Related Desynchronization (ERD). More negative values indicate greater Beta-band ERD at post-intervention.
Time Frame: Baseline to approximately 4 weeks
Population: Subjects were removed from analysis if their data was too noisy from excessive coughing or moving around.
Measure: Mean (Standard Deviation); unit: microvolts squared
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 7 | 5 | 7 | 5
microvolts squared | -3.8 (2.6) | -2.6 (3.1) | -3.6 (6.2) | -0.2 (4.6)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Test of between-subjects effects; Test type: Superiority; p = .564, ANOVA; P-value indicates the interaction term

10. Secondary Outcome: Attention & Smoking Cue Exposure Task (ASCET)
Description: Post minus Pre-intervention difference in Reaction time between smoking and neutral images presented with the ASCET task. A negative RT indicates improvement.
Time Frame: Baseline to approximately 4 weeks
Population: The baseline data for one subject in CR + tDCS did not save.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 6 | 6 | 9 | 8
milliseconds | -21.9 (19.6) | -21.7 (23.0) | -10.5 (23.3) | -8.6 (32.8)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Tests of between-subjects effects; Test type: Superiority; p = .998, ANOVA; p-value indicates the interaction term

11. Secondary Outcome: Total Number of Puffs
Description: Change in number of puffs on cigarettes assessment during smoking topography measurement during the cue reactivity task. Number of puffs was assessed during pre-training cue reactivity and again during post-training cue reactivity.
Time Frame: Baseline to approximately 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
Number analyzed (Participants) | 6 | 4 | 7 | 8
puffs | -7.3 (11.3) | 0.8 (7.8) | -2.0 (11.1) | 2.0 (15.7)
Statistical Analysis 1: Comparison: CR + tDCS vs CR + Sham tDCS vs Control CR + tDCS vs Control CR + Sham tDCS; Tests of between-subjecs effects; Test type: Superiority; p = .348, ANOVA; P-value indicates the interaction term

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events from the time they completed informed content to the end of their participation in the study, which was approximately 4 weeks.
Arm/Group | CR + tDCS | CR + Sham tDCS | Control CR + tDCS | Control CR + Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 0/6 | 0/12 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR + tDCS (N=10) | CR + Sham tDCS (N=6) | Control CR + tDCS (N=12) | Control CR + Sham tDCS (N=11)
Illness not related to study participation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant was hospitalized Briefly due to illness not related to study participation.

LIMITATIONS AND CAVEATS:
Study was unexpectedly shut down prior to completing recruitment due to COVID-19 protocols.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT03588728/Prot_SAP_000.pdf